CLINICAL TRIAL: NCT02999906
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Compare the Efficacy and Safety of Triple Therapy (Oral Treprostinil, Ambrisentan, and Tadalafil) With Dual Therapy (Ambrisentan, Tadalafil, and Placebo) in Subjects With Pulmonary Arterial Hypertension
Brief Title: Study to Compare Triple Therapy (Oral Treprostinil, Ambrisentan, and Tadalafil) With Dual Therapy (Ambrisentan, Tadalafil, and Placebo) in Subjects With Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: For business reasons.
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-PH-313
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Oral Treprostinil; dual therapy; 6 Minute Walk Test
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo (sugar pill)
  Interventions: Drug: Placebo
- Active (Active Comparator): Oral treprostinil sustained release tablet
  Interventions: Drug: Oral Treprostinil

INTERVENTIONS:
Drug: Oral Treprostinil — Sustained release oral tablets for three times daily administration
  Other Names: treprostinil diethanolamine
  Arms: Active
Drug: Placebo — Placebo (sugar pill) for three times daily oral administration
  Other Names: matching placebo (sugar pill)
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized (2:1 oral treprostinil: placebo), double-blind, placebo-controlled study in subjects with Pulmonary Arterial Hypertension (PAH) who are currently receiving background dual therapy (ambrisentan, tadalafil) for at least 30 days at randomization for their PAH. Once randomized, subjects will return for 5 study visits up to Week 28 during the blinded period. After the Week 28 Visit, eligible subjects will transition to the open-label period of the study for up to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 79 years of age, inclusive
2. PAH that is idiopathic / heritable, PAH associated with connective tissue disease, HIV infection, repaired congenital systemic-to-pulmonary shunts (repaired > 1 year), or appetite suppressant / toxin use
3. Receiving dual therapy (ambrisentan and tadalafil)
4. Previous testing (e.g. right heart catheterization, echocardiography) consistent with diagnosis of PAH

Exclusion Criteria:

1. Nursing or pregnant
2. PAH due to conditions other than noted in the above inclusion criteria
3. Received PAH-specific drug therapy for >2 years
4. History of uncontrolled sleep apnea, severe liver disease, severe renal impairment, left sided heart disease, uncontrolled systemic hypertension
5. Participated in an investigational drug or device study within 90 days prior to signing consent.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Distance (6MWD) | Baseline to Week 28

SECONDARY OUTCOMES:
Compare the effects of triple therapy versus dual therapy on the time to clinical worsening | Baseline to Week 28
  clinical worsening is defined by 1 of the following:
  * Death (all causes)
  * Hospitalization due to worsening PAH
  * Initiation of long-term parenteral therapy
  * Disease progression
  * Unsatisfactory long-term clinical response
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) concentrations From Baseline to Week 28 | Baseline to week 28
  The level of this biomarker of the (NT-proBNP) serum concentration will be assessed to compare the severity of heart failure at Baseline and Week 28.
Number of Participants with a Change From Baseline World Health Organization (WHO) Functional Classification at Week 28. | Baseline to week 28
  The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
Change in Quality of Life (QoL) Assessment: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) From Baseline to Week 28. | Baseline to week 28
  The CAMPHOR is a health related quality of life instrument validated for pulmonary hypertension that assesses impairment (symptoms), disability (activities) and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 025; high scores indicate more symptoms), Activity (Score 030; low score indicates good functioning) and Quality of Life (025; high scores indicate poor QoL). The sum of these scores equates to the Total score (080). In the CAMPHOR scores, lower scores indicate improvements.

IPD SHARING:
Plan to Share IPD: No